CLINICAL TRIAL: NCT04612075
Title: The EMINENCE Study - PET/MR Imaging of Head Neck Cancer
Acronym: EMINENCE
Status: Recruiting | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); University Hospital of North Norway (Other); University of Bergen (Other)
Responsible Party: Sponsor
Other Study IDs: 64744
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Neoplasms
Keywords: Diagnostic Imaging; Functional Imaging; Nuclear magnetic Resonance Imaging; Positron-Emission Tomography; Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- All patients referred to fast track clinical pathway for HNC cancer: MRI as part of staging, including a 5-minute additional sequence.
- Patients with locally advanced HNC: FDG-PET/MRI
  Interventions: Diagnostic Test: FDG-PET/MRI

INTERVENTIONS:
Diagnostic Test: FDG-PET/MRI — Performed at baseline, interim and at 12-16 weeks post radiotherapy.
  Groups: Patients with locally advanced HNC

SUMMARY:
Head and neck cancers (HNC) often receive radiotherapy as part of their treatment. However, unacceptable failure rates and severe side effects remain a challenge. The improvements in radiotherapy are closely related to improvements in medical imaging. Functional imaging, where intratumoural characteristics such as tumour oxygenation, metabolism, and blood vessel function can be quantified, offers possibilities to personalize the radiotherapy. In this study we will establish the clinical workflow for PET- and MRI-based radiotherapy in HNC by acquiring images prior to and during radiotherapy to develop new concepts for image-based biologically adaptive radiotherapy, both based on photon-based radiotherapy and also proton therapy, which soon will be available for cancer patients in Norway. The investigators aim to contribute towards further developments of personalised high-precision radiotherapy for HNC patients resulting in improved outcome, reduced side-effects and better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to give full written consent according to the protocol approved by the Regional Ethics Committee
* histologically confirmed squamous cell carcinoma in the head neck region (pharynx, larynx, oral cavity or sinonasal area)
* locally advanced disease without sign of dissemination (T3/T4 and/or N1-3, M0) on diagnostic imaging
* scheduled for definitive radiotherapy with curative intent with or without concomitant chemotherapy
* adequate renal function: Creatinine clearance ≥ 60 ml/minute
* lymph node metastasis from cancer of unknown primary of the upper neck (i.e. level II-III) were PET/CT is negative outside the head-neck region can be considered for inclusion at the discretion of the study investigators.

Exclusion Criteria:

* general contraindications for MRI (pacemaker, aneurysm clips, any form of metal in the body, severe claustrophobia)
* serious comorbidity (including previous or othe cancer) that in the opinion of the investigator would compromise the patient's ability to complete the study of interfere with the evaluation of the study objectives (e.g. poorly controlled diabetes mellitus)
* histologically confirmed SCC of same or other origin within the last five years
* patient wants to withdraw for any reason during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population 1 consists of all patients who are referred to the "fast track" clinical pathway for HNC at St. Olavs hospital, approximately 130 patients per year for three years. Out of these, 60 patients are defined as study population 2, due to locally advanced head and neck cancer (HNC) of squamous cell histology scheduled for definitive (chemo)radiotherapy with curative intent.
Sampling Method: Non-Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Population 1: Predict overall survival five years after treatment | Five years after treatment
  For study population one, the primary study objective is to explore the potential of functional MR imaging parameters in predicting overall survival in head and neck cancer (HNC) five years after treatment.
Population 2: Response three months after treatment | Three months after treatment
  For study population two, the primary objective is response three months after treatment.

SECONDARY OUTCOMES:
Populations 1 and 2: Time to local relapse and time to distant metastasis | Five years after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Torstein Baade Rø, md phd, Study Director — Norwegian University of Science and Technology, IKOM; Arne Solberg, md phd, Study Director — St Olavs Hospital, Dept Oncology; Erik Wahlström, phd, Study Director — Norwegian University of Science and Technology, Institute for Fysikk
Locations (2):
- Norway (2):
  - University Hospital of North Norway, Tromsø
  - St Olavs Hospital, Department of Oncology, Trondheim